CLINICAL TRIAL: NCT06350461
Title: A Master Protocol to Test the Impact of Discontinuing Chronic Therapies in People With Cystic Fibrosis on Highly Effective CFTR Modulator Therapy - Hypertonic Saline
Brief Title: Impact of Discontinuing Hypertonic Saline in People With CF on Highly Effective CFTR Modulators- A SIMPLIFY Sub-Study
Acronym: SIMPLIFY-HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Dartmouth-Hitchcock Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor of Pediatrics, Division of Pulmonary and Sleep Medicine, University of Washington School of Medicine Adjunct Professor, Biostatistics, University of Washington School of Medicine Co-Executive Director, Cystic Fibrosis Therapeutics Development, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIMPLIFY-IP-19 HS
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF; Withdrawal; ETI; hypertonic saline; discontinue
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-Discontinue (Experimental): Discontinuation of current hypertonic saline (HS) therapy
  Interventions: Other: Discontinuation of hypertonic saline (HS)
- HS-Continue (Active Comparator): Continuation of current hypertonic saline (HS) therapy
  Interventions: Other: Continuation of hypertonic saline (HS)

INTERVENTIONS:
Other: Discontinuation of hypertonic saline (HS) — Discontinuation of current hypertonic saline (HS) therapy during 6-week study period.
  Arms: HS-Discontinue
Other: Continuation of hypertonic saline (HS) — Continuation of current hypertonic saline (HS) therapy during 6-week study period. Therapy is taken at least once daily according to each participant's pre-existing, clinically prescribed regimen (e.g., daily, twice daily). The concentration of HS is according to clinical prescription (e.g., 7% sodium chloride or 3.5% sodium chloride) and at least 3%.
  Arms: HS-Continue

SUMMARY:
Despite the increasingly common use of cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapies in treating cystic fibrosis (CF), it is still largely unknown whether or not other chronic therapies can be safely stopped. This SIMPLIFY sub-study is being done to test whether or not it is safe to stop taking inhaled hypertonic saline in those people that are also taking elexacaftor/tezacaftor/ivacaftor (ETI).

ETI is a combination CFTR modulator therapy that was approved by the Food and Drug Administration for people with CF who have at least one F508del mutation. The three drugs that make up ETI work together to allow many more chloride ions to move into and out of the cells, improving the balance of salt and water in the lungs. These changes result in better clearance of mucus from the lungs and improvements in lung function.

Inhaled hypertonic saline (HS) also improves clearance of mucus from the lungs to support lung function and has been available to people with CF for many years. HS is considered to be relatively burdensome and it is not known whether HS can improve or maintain lung function above what is already gained through ETI use.

The goal of this SIMPLIFY sub-study is to get information about whether or not it is safe to stop hypertonic saline by testing if there is a change in lung function in participants with cystic fibrosis (CF) who are assigned to stop taking HS as compared to those who are assigned to keep taking HS while continuing to take ETI.

This is a sub study of master protocol SIMPLIFY-IP-19, NCT04378153.

The sub study investigating the impact of discontinuing and continuing dornase alfa is registered under NCTXXXXXXX (will add once available).

DETAILED DESCRIPTION:
This SIMPLIFY sub-study (Hypertonic Saline (HS) Trial) is designed to evaluate the effects of discontinuing HS in people with cystic fibrosis (CF) age 12 and older currently taking the highly effective modulator elexacaftor/tezacaftor/ivacaftor (ETI). This is an open label two-arm randomized non-inferiority trial consisting of a 2-week screening period, randomization to continue or discontinue hypertonic saline, followed by a 6-week study period. Participants at trial entry will be randomized 1:1 to either continue or discontinue their HS therapy.

Clinical outcomes (forced expiratory volume in 1 second [FEV1], antibiotic use, pulmonary exacerbations, and patient reported outcomes), safety (adverse events) and patient reported outcomes to evaluate respiratory symptoms and the participant's perception of how stopping HS would impact their daily life will be evaluated in all subjects. Additionally, a subset of participants at selected study sites will participate in Multiple Breath Washout (MBW) to evaluate changes in lung clearance index (LCI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF.
* Age ≥ 12 years at the Screening Visit.
* Forced expiratory volume in 1 second (FEV1) ≥ 70 % predicted at the Screening Visit if < 18 years old, and ≥ 60 % predicted at Screening Visit if ≥ 18 years old.
* Clinically stable with no significant changes in health status within the 7 days prior to and including the Screening Visit.
* Current treatment with elexacaftor/tezacaftor/ivacaftor (ETI) for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the duration of the study.
* Currently taking hypertonic saline (at least 3%) for at least the 90 days prior to and including the Screening Visit and willing to continue daily use for the 2-week screening period.

Exclusion Criteria:

* Active smoking or vaping.
* Use of an investigational drug within 28 days prior to and including the Screening Visit.
* Changes to chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, aztreonam lysine) within 28 days prior to and including the Screening Visit. This includes new airway clearance routines.
* Acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within 7 days prior to and including the Screening Visit.
* Chronic use of systemic corticosteroids at a dose equivalent to ≥ 10mg per day of prednisone within 28 days prior to and including the Screening Visit.
* Antibiotic treatment for nontuberculous mycobacteria (NTM) within 28 days prior to and including the Screening Visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Mayer-Hamblett, PhD, Principal Investigator — University of Washington/Seattle Children's; Alex Gifford, MD, FCCP, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (81):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - CHOC Children's Hospital, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital and Health Center at the University of California San Diego, San Diego, California
  - University of California, San Francisco - Adult Center, San Francisco, California
  - University of California, San Francisco - Peds Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Tulane University, Metairie, Louisiana
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Wayne State University Harper University Hospital, Detroit, Michigan
  - Corewell Health Helen DeVos, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Eatontown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Lenox Hill Hospital Cystic Fibrosis Center, New York, New York
  - Columbia University Cystic Fibrosis Program, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cystic Fibrosis Program, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Primary Children's Cystic Fibrosis Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Medical Group, Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HS-Discontinue | HS-Continue
Started | 184 | 186
Completed | 181 | 183
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Primary analyses were done on the per-protocol (PP) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | HS-Discontinue | HS-Continue | Total
Number analyzed (Participants) | 133 | 140 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (11.06) | 23.5 (11.34) | 22.7 (11.22)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution (years): >=12 to 18 | 68 | 64 | 132
  Age Distribution (years): >=18 to <24 | 24 | 28 | 52
  Age Distribution (years): >=24 to <30 | 22 | 15 | 37
  Age Distribution (years): >=30 | 19 | 33 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 128
  Male | 68 | 77 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 122 | 134 | 256
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 128 | 136 | 264
  Race: Black or African American | 2 | 1 | 3
  Race: Asian | 0 | 0 | 0
  Race: American Indian or Alaskan Native | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other, More than one Race, or Unknown/Not Reported | 3 | 3 | 6
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants]
  F508 Homozygous | 82 | 84 | 166
  F508 Heterozygous | 51 | 53 | 104
  Other or Unknown | 0 | 3 | 3
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Liters] | 3.4 (0.91) | 3.4 (0.89) | 3.4 (0.90)
FEV1 (% Predicted) Distribution [Count of Participants; unit: Participants] — FEV1 % predicted is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  Participants
    <60 | 1 | 1 | 2
    >=60 to <70 | 9 | 10 | 19
    >=70 to <90 | 32 | 37 | 69
    >=90 to <100 | 31 | 26 | 57
    >=100 | 60 | 66 | 126
FEV1 (% Predicted) [Mean (Standard Deviation); unit: Percent of Predicted] — FEV1 % predicted is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  Percent of Predicted | 97.6 (17.55) | 96.8 (17.30) | 97.2 (17.40)
Current Dornase Alfa Use [Count of Participants; unit: Participants] — Use as reported at screening prior to randomization
  Participants | 111 | 120 | 231
Current Airway Clearance Use [Count of Participants; unit: Participants] — Includes airway clearance by route chest PT/vest.
  Participants | 127 | 132 | 259
Previous Enrollment in SIMPLIFY-DA Study [Count of Participants; unit: Participants]
  Yes | 42 | 45 | 87
  No | 91 | 95 | 186

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in FEV1 % Predicted From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week 0 to Week 6.
Time Frame: Week 0 to Week 6
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: FEV1 % predicted
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 133 | 140
FEV1 % predicted | -0.2 (4.10) | 0.1 (3.64)
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; The non-inferiority test was a priori designed to be conducted on the per-protocol (PP) population; Test type: Non-Inferiority — The non-inferiority margin is -3; p < 0.0001, ANOVA — One-sided test for non-inferiority; Adjusted for four dichotomous randomization strata; Median Difference (Final Values) = -0.324, 95% CI 2-sided [-1.3 to 0.6] — Direction of difference is Discontinue - Continue

2. Secondary Outcome: Absolute Change in LCI 2.5 From Baseline to Week 6
Description: Difference between study arms (discontinue - continue) in the absolute change in LCI 2.5 (Lung Clearance Index) from Baseline (Week 0, if available, or else Week -2) to Week 6. LCI 2.5 is the number of times the volume in the lungs needs to turn over to expel an inert gas. A higher value of LCI 2.5 indicates poorer lung function.
Time Frame: Baseline (Week 0 or Week -2) to Week 6
Population: Participants in the per-protocol (PP) population with an acceptable LCI 2.5 measurement at baseline and at Week 6.
Measure: Mean (Standard Deviation); unit: number of lung volume turnovers
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 31 | 28
number of lung volume turnovers | 0.1 (0.72) | 0.1 (0.73)
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Test type: Superiority; p = 0.733, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.4 to 0.4] — Direction of difference is Discontinue - Continue

3. Secondary Outcome: Absolute Change in Respiratory Symptoms, as Measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CRISS) From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the absolute change in respiratory symptoms, as measured by the CF Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CRISS) from Week 0 to Week 6. The Cystic Fibrosis Respiratory Symptoms Daily Diary (CFRSD) asks a participant to state the extent of their 8 respiratory symptoms: difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present 'a great deal' or 'extremely'. A summed score (range from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100, where the lowest scores indicate improvement of symptoms. Calculation of a score requires responses for at least 7 out of 8 symptoms.
Time Frame: Week 0 to Week 6
Population: Participants in the per-protocol (PP) population with a CRISS score at Week 0 and Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 132 | 140
score on a scale | -1.4 (11.02) | 0.2 (9.73)
Statistical Analysis 1: Comparison: HS-Discontinue; Test type: Superiority; p = 0.226, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-4.1 to 0.9] — Direction of difference is Discontinue - Continue

4. Secondary Outcome: Absolute Change in Respiratory Symptoms, as Measured by CFQ-R Respiratory Domain From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the absolute change in respiratory symptoms, as measured by the Cystic Fibrosis Questionnaire-Revised Respiratory Domain Score from Week 0 to Week 6. The Cystic Fibrosis Questionnaire - Revised asks participants 6 questions related to respiratory symptoms which are each assigned a score 1-4. The Respiratory Domain Scaled Score is calculated as follows: 100*[{sum of responses}/{number of responses}-1]/3 only if number of responses ≥ 3; otherwise the score is set to missing. The scaled score ranges from 0 to 100 where higher scores indicate improvement of symptoms.
Time Frame: Week 0 to Week 6
Population: Participants in the per-protocol (PP) population with a score at Week 0 and at Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 133 | 140
score on a scale | 0.7 (9.56) | 0.5 (6.35)
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Test type: Superiority; p = 0.857, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-1.8 to 2.1] — Direction of the difference is Discontinue - Continue

5. Secondary Outcome: Absolute Change in FEV1 % Predicted From Week -2 to Week 0
Description: Difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week -2 to Week 0.
Time Frame: Week -2 to Week 0
Population: Per-protocol (PP) population
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 133 | 140
% predicted | 0.2 (3.63) | -0.4 (3.86)
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.25 to 1.54] — Direction of the difference is Discontinue - Continue

6. Secondary Outcome: Absolute Change in FEV1 % Predicted From Week 0 to Week 2
Description: Difference between study arms (discontinue - continue) in the absolute change in FEV1 % predicted from Week 0 to Week 2.
Time Frame: Week 0 to Week 2
Population: Participants in the per-protocol (PP) population with FEV1 measurements at Week 0 and at Week 2
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 128 | 138
% predicted | 0.3 (3.66) | 0.6 (2.94)
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Test type: Superiority; p = 0.56, t-test, 2 sided; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.04 to 0.57] — Direction of the difference is Discontinue - Continue

7. Secondary Outcome: Number and Percent of Participants Initiating Acute Antibiotics From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of subjects initiating acute oral, inhaled or intravenous antibiotics from Week 0 to Week 6. Includes antibiotics initiated for respiratory indications; excludes those taken as part of a chronic cycled regimen or for a UTI, skin infection, etc.
Time Frame: Week 0 to Week 6
Population: Intent to treat (ITT) population of all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
Participants | 11 | 9
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Null hypothesis: proportion of participants initiating acute antibiotics is the same in the Discontinue and Continue arms; Test type: Superiority; p = 0.653, Fisher Exact; Difference in % Participants = 1.1, 95% CI 2-sided [-3.7 to 6.1] — Confidence interval calculated using the Newcombe-Wilson method without continuity correction. Direction of difference is Discontinue - Continue

8. Secondary Outcome: Number and Percent of Participants Hospitalized From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of subjects hospitalized from Week 0 to Week 6.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
Participants | 2 | 1
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Null hypothesis: proportion of participants with at least one hospitalization is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.622, Fisher Exact; Difference in % Participants = 0.5, 95% CI 2-sided [-2.0 to 3.4] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Number and Percent of Participants Experiencing Pulmonary Exacerbations From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of subjects experiencing a pulmonary exacerbation from Week 0 to Week 6. Pulmonary exacerbations defined using Fuchs criteria.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
Participants | 1 | 3
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Null hypothesis: proportion of participants with at least one protocol-defined pulmonary exacerbation is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.623, Fisher Exact; Difference in % Participants = -1.1, 95% CI 2-sided [-4.1 to 1.6] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Number and Percent of Participants Experiencing Adverse Events (AEs) From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of participants with at least one AE from Week 0 to Week 6. Includes serious and non-serious AEs.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
Participants | 65 | 44
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Null hypothesis: proportion of participants with at least one AE is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.0165, Fisher Exact; Difference in % Participants = 11.7, 95% CI 2-sided [2.4 to 20.7] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Rate of Adverse Events (AEs) From Week 0 to Week 6 Therapy Arms
Description: Comparison of study arms (discontinue/continue) in the rate of AE occurrence (number of events divided by total follow-up weeks in each arm) from Week 0 to Week 6. Includes serious and non-serious AEs.
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Number; unit: events per week
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
events per week | 0.086 | 0.067
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Rate ratio, confidence interval, and p-value calculated using Poisson Regression with an offset for the log of follow-up time in weeks. The total number of follow-up weeks in the HS-discontinue and HS-continue arms are 1135.7 and 1163.9 weeks, respectively. Ratio is Discontinue / Continue; Test type: Superiority; p = 0.0958, Poisson Regression; Rate Ratio = 1.29, 95% CI 2-sided [0.96 to 1.74]

12. Secondary Outcome: Number and Percent of Participants With Temporary or Permanent Changes From Assigned Therapy Regimen Due to Adverse Event From Week 0 to Week 6
Description: Difference between study arms (discontinue - continue) in the percent of subjects temporarily or permanently changing their assigned therapy regimen due to an adverse event Week 0 to Week 6
Time Frame: Week 0 to Week 6
Population: Intent-to-treat (ITT) population of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | HS-Discontinue | HS-Continue
Number analyzed (Participants) | 184 | 186
Participants | 5 | 1
Statistical Analysis 1: Comparison: HS-Discontinue vs HS-Continue; Null hypothesis: proportion of participants changing assigned regimen is the same in Discontinue and Continue arms; Test type: Superiority; p = 0.1215, Fisher Exact; Difference in % Participants = 2.17, 95% CI 2-sided [-0.7 to 5.7] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: From randomization (Week 0) up to last study visit (Week 6), i.e., 6 weeks.
Arm/Group | HS-Discontinue | HS-Continue
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/186
Serious Adverse Events (participants affected / at risk) | 2/184 | 1/186
Other Adverse Events (participants affected / at risk) | 5/184 | 10/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HS-Discontinue (N=184) | HS-Continue (N=186)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HS-Discontinue (N=184) | HS-Continue (N=186)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT06350461/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT06350461/SAP_001.pdf